CLINICAL TRIAL: NCT04407871
Title: Acupuncture and Chinese Herbal Medicine to Improve Live Birth Rate of in Vitro Fertilization - A Randomized Controlled Trial (IVFAct)
Brief Title: Acupuncture and Chinese Herbal Medicine to Improve Live Birth Rate of in Vitro Fertilization (IVFAct)
Acronym: IVFAct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Director of Obstetrics and Gynecology Department, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVFAct
Record Dates: First submitted 2020-05-18; First posted 2020-05-29 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: In Vitro Fertilization
Keywords: In Vitro Fertilization; Chinese Herbal Medicine; Acupuncture; Live Birth
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- acupuncture and CHM (Experimental): Women will receive acupuncture three times a week 4 weeks prior to ovarian stimulation for IVF and during ovarian stimulation, and before and after embryo transfer (ET). They will also take CHM daily 4 weeks prior to IVF till the day of serum hCG testing. If the hCG testing is positive and a viable pregnancy is confirmed by transvaginal ultrasound, CHM will be continued till 8 weeks of gestation. If the hCG testing is negative or spontaneous miscarriage is confirmed, the drug treatment will be stopped.
  Interventions: Other: Acupuncture and Chinese Herbal Medicine
- acupuncture and placebo CHM (Placebo Comparator): Women will receive acupuncture three times a week 4 weeks prior to ovarian stimulation for IVF and during ovarian stimulation, and before and after ET. They will also take placebo CHM daily 4 weeks prior to IVF till the day of serum hCG testing. If the hCG testing is positive and a viable pregnancy is confirmed by transvaginal ultrasound, placebo CHM will be continued till 8 weeks of gestation. If the hCG testing is negative or spontaneous miscarriage is confirmed, the drug treatment will be stopped.
  Interventions: Other: Acupuncture and Chinese Herbal Medicine
- control acupuncture and CHM (Placebo Comparator): Women will receive control acupuncture three times a week 4 weeks prior to ovarian stimulation for IVF and during ovarian stimulation, and before and after ET. They will also take CHM daily 4 weeks prior to IVF till the day of serum hCG testing. If the hCG testing is positive and a viable pregnancy is confirmed by transvaginal ultrasound, CHM will be continued till 8 weeks of gestation. If the hCG testing is negative or spontaneous miscarriage is confirmed, the drug treatment will be stopped.
  Interventions: Other: Acupuncture and Chinese Herbal Medicine
- control acupuncture and placebo CHM (Placebo Comparator): Women will receive control acupuncture three times a week 4 weeks prior to ovarian stimulation for IVF and during ovarian stimulation, and before and after ET. They will also take placebo CHM daily 4 weeks prior to IVF till the day of serum hCG testing. If the hCG testing is positive and a viable pregnancy is confirmed by transvaginal ultrasound, placebo CHM will be continued till 8 weeks of gestation. If the hCG testing is negative or spontaneous miscarriage is confirmed, the drug treatment will be stopped.
  Interventions: Other: Acupuncture and Chinese Herbal Medicine

INTERVENTIONS:
Other: Acupuncture and Chinese Herbal Medicine — 1) acupuncture and CHM, 2) acupuncture and placebo CHM, 3) control acupuncture and CHM or 4) control acupuncture and placebo CHM by an interactive online computer program in a central office. Using a 1:1:1:1 treatment ratio, there will be 682 women assigned to each treatment group.

SUMMARY:
The most successful treatment for infertility is in vitro fertilization (IVF), but less than 10% of infertile couples undergo IVF because of the high cost and relatively low success rate. Many patients have tried complementary and alternative medical treatments as an adjuvant therapy to improve their IVF success. Acupuncture given 2-4 times around the day of embryo transfer has not been shown to improve the IVF live birth rate. Chinese Herbal Medicine (CHM) may improve the IVF pregnancy rates, but the evidence so far is inconclusive because of high risks of bias in these studies.

The objective of this multi-centre double blind randomized trial is to evaluate the efficacy of acupuncture with or without CHM on the live birth of IVF. The randomization process will be coordinated through a central mechanism. A total of 2,728 subjects will be randomized in 1:1:1:1 ratio in to one of the four treatment arms: 1) acupuncture and CHM, 2) acupuncture and placebo CHM, 3) control acupuncture and CHM or 4) control acupuncture and placebo CHM. Women will receive acupuncture or control acupuncture three times a week 4 weeks prior to IVF during ovarian stimulation, and before and after the embryo transfer. They will also take CHM or placebo CHM daily 4 weeks prior to IVF till a negative pregnancy test or till 8 weeks of gestation if pregnant.

DETAILED DESCRIPTION:
The objective of this multi-centre double blind randomized trial is to evaluate the efficacy of acupuncture with or without CHM on the live birth of IVF. The randomization process will be coordinated through a central mechanism. A total of 2,728 subjects will be randomized in 1:1:1:1 ratio in to one of the four treatment arms: 1) acupuncture and CHM, 2) acupuncture and placebo CHM, 3) control acupuncture and CHM or 4) control acupuncture and placebo CHM. Women will receive acupuncture or control acupuncture three times a week 4 weeks prior to IVF during ovarian stimulation, and before and after the embryo transfer. They will also take CHM or placebo CHM daily 4 weeks prior to IVF till a negative pregnancy test or till 8 weeks of gestation if pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥20 to ≤40 years of age
2. Indications for IVF
3. Duration of infertility >1 year
4. Undergoing IVF with an intention of fresh ET on day 3 or 5.

Exclusion Criteria:

1. Women with an intention to replace frozen embryos only.
2. Preimplantation genetic testing
3. History of recurrent miscarriages defined as having three consecutive miscarriages.
4. Having acupuncture or CHM for infertility within 3 months prior the IVF
5. Women with abnormal liver or renal function tests

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Undergoing IVF
Enrollment: 2728 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth | ≥20 weeks of gestation
  Live birth defined as a delivery ≥20weeks gestation per transfer in the stimulated IVF cycles or in the first frozen-thawed embryo transfer cycle in those with elective freezing of all embryos

SECONDARY OUTCOMES:
Embryo quality: embryo scoring standard | On the third day after egg retrieval and before embryo transfer
  Embryo quality is judged by embryo scoring standard
Miscarriage rate | ≤42 weeks of gestation
  Cumulative miscarriage rate
Implantation rate | 2 weeks after embryo transfer
  Cumulative implantation rate
Positive serum human chorionic gonadotropin (hCG) level | 2 weeks after embryo transfer
  Positive serum hCG level 2 weeks after embryo transfer
Ongoing pregnancy rate | ≥8 weeks
  Cumulative ongoing pregnancy rate
Multiple pregnancy rate | ≥2 weeks after embryo transfer
  Cumulative multiple pregnancy rate
Ectopic pregnancy rate | ≥2 weeks after embryo transfer
  Cumulative ectopic pregnancy rate
Cumulative live birth rate | within 6 months after randomization
  Cumulative live birth rate
Changes in markers of stress, anxiety | ≤8 weeks of gestation
  To elucidate the anxiety level as measured with serum cortisol concentration and Stait-Trait Anxiety Inventory (STAI)
Health related quality of life(HRQoL) | ≤8 weeks of gestation
  To determine women's health related quality of life (HRQoL) by short-form 36 (SF36)
Patient acceptability: acupuncture trust score | On the day of embryo transfer
  Patient acceptability of acupuncture to be measured by acupuncture trust score
Side effects | ≤ 8 weeks of gestation
  Side effects
Congenital abnormalities | at 6 weeks postpartum
  Judging by prenatal ultrasound and postnatal physical examination
Pregnancy complications | ≤42 weeks of gestation
  Complications of Pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoke Wu, Ph.D, Study Chair — First Affiliated Hospital in Heilongjiang University of Chinese Medicine
Locations (12):
- China (12):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - Huaian Maternal and Child Health Hospital, Huai'an, Jiangsu
  - The First Affiliated Hospital of Nanjing University Medical School (Nanjing Drum Tower Hospital), Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Dalian Municipal Women and Children's Medical Center, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Xibei Women and Children's Hospital, Xi’an, Shanxi
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Subject's privacy is protected undoubtedly at the time of the informed consent signing